CLINICAL TRIAL: NCT03982979
Title: MOMENTUM 3 Pivotal Cohort Extended Follow-up Post-Approval Study
Brief Title: MOMENTUM 3 Pivotal Cohort Extended Follow-up PAS
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10273
Record Dates: First submitted 2019-05-16; First posted 2019-06-12 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Advanced Refractory Left Ventricular Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: HM3 LVAS — HeartMate® 3 (HM3) Left Ventricular Assist System (LVAS)

SUMMARY:
The study will be a prospective, multi-center, non-blinded, controlled study, intended to evaluate the extended use of the HM3 LVAS compared to the HMII LVAS in those patients that are ongoing at the 2-year follow-up in the MOMENTUM 3 IDE trial. A total of 1028 subjects were enrolled in the MOMENTUM 3 IDE trial. Approximately 533 subjects were ongoing support at the 2-year follow-up and are eligible for enrollment in this PAS. This study will be conducted at sites that participated in the MOMENTUM 3 IDE trial which will include up to 69 centers in the United States.

DETAILED DESCRIPTION:
Subjects on LVAD support after the MOMENTUM 3 IDE trial 2-year follow-up visit can be enrolled after providing consent to extended follow-up. They will be followed to 5 years post-implant or outcome (transplant, explant or death), whichever occurs first.

Subjects who have been transplanted, their device exchanged to another pump other than a HM II or HM3, or explanted after the MOMENTUM 3 IDE trial 2-year follow-up but prior to providing consent for this PAS can also be enrolled. Data between the 2-year follow-up visit and the date of pump exchange, explant, or transplant will be retrospectively collected.

Once enrolled, if subjects receive a device exchange to any device other than HM II or HM3, at any time during the study, they will be withdrawn from the study and will not be followed.

In the event that a subject expired prior to providing consent, IRB approval will be obtained to collect the date and cause of death.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legal representative has signed Informed Consent Form (ICF)
* Subject was enrolled in the MOMENTUM 3 IDE trial and was ongoing at the 2-year follow-up visit

Exclusion Criteria:

* Subject or legal representative does not consent to extended data collection after the MOMENTUM 3 IDE trial 2-year follow-up visit

Special Circumstance:

* Sites with patients who expired after the MOMENTUM 3 IDE trial 2-year follow-up visit but prior to signing the ICF for this PAS will obtain IRB approval to collect only the date and cause of death

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: As part of the PAS requirement, this study will consent male and female subjects with advanced refractory left ventricular heart failure who were implanted with the HM3 or HMII LVAS in the MOMENTUM 3 IDE trial and are ongoing at the 2-year follow up. Subjects must meet all eligibility criteria and provide written informed consent prior to conducting any investigation-specific procedures not considered standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Survival | up to 5 years post-implant
  Composite of Survival to transplant, recovery, or LVAD support free of debilitating stroke (Modified Rankin Score > 3) or reoperation to replace the pump
Subject outcomes and survival | up to 5 years post-implant
  Subject outcomes and survival which includes death, transplant, explant, or a pump exchange to any device other than HM II or HM3
Bleeding (including GI bleeding) | up to 5 years post-implant
  Frequency and incidence of bleeding (including GI bleeding)
Major infection | up to 5 years post-implant
  Frequency and incidence of major infection
Hemolysis | up to 5 years post-implant
  Frequency and incidence of hemolysis
Device thrombosis | up to 5 years post-implant
  Frequency and incidence of device thrombosis
Neurological dysfunction | up to 5 years post-implant
  Frequency and incidence of neurological dysfunction
Device related SAEs | up to 5 years post-implant
  Frequency and incidence of device related SAEs
NYHA | up to 5 years post-implant
  New York Heart Association (NYHA) classification
6MWD | up to 5 years post-implant
  Six-minute walk distance (6MWD)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elena Brett, PhD, Study Director — Abbott
Locations (1):
- Abbott, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nayak A, Hall SA, Uriel N, Goldstein DJ, Cleveland JC Jr, Cowger JA, Salerno CT, Naka Y, Horstmanshof D, Crandall D, Wang A, Mehra MR. Predictors of 5-Year Mortality in Patients Managed With a Magnetically Levitated Left Ventricular Assist Device. J Am Coll Cardiol. 2023 Aug 29;82(9):771-781. doi: 10.1016/j.jacc.2023.05.066. PMID 37612008
- [Derived] Mehra MR, Goldstein DJ, Cleveland JC, Cowger JA, Hall S, Salerno CT, Naka Y, Horstmanshof D, Chuang J, Wang A, Uriel N. Five-Year Outcomes in Patients With Fully Magnetically Levitated vs Axial-Flow Left Ventricular Assist Devices in the MOMENTUM 3 Randomized Trial. JAMA. 2022 Sep 27;328(12):1233-1242. doi: 10.1001/jama.2022.16197. PMID 36074476